CLINICAL TRIAL: NCT00090246
Title: A Randomized, Double-Blind, Active Comparator-Controlled, Parallel-Group Study, Conducted Under In-House Blinding Conditions, to Examine the Safety, Tolerability, and Efficacy of 2 Doses of Aprepitant for the Prevention of Postoperative Nausea and Vomiting
Brief Title: 2 Doses of an Approved Drug Being Studied for a New Indication for the Prevention of Postoperative Nausea and Vomiting (0869-091)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0869-091; 2004_014
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0869, aprepitant
Drug: Comparator: ondansetron IV

SUMMARY:
The purpose of this study is to assess the safety and efficacy of 2 doses of an approved drug for a new indication in the prevention of postoperative nausea and vomiting in patients receiving general anesthesia for open abdominal surgery requiring overnight hospital stay.

DETAILED DESCRIPTION:
The duration of treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient is scheduled to undergo open abdominal surgery requiring overnight hospital stay (24-hour hospital stay after end of surgery).
* Patient is scheduled to receive general anesthesia.
* Patient is scheduled to receive postoperative opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Actual)
Dates: Start 2004-05-13 (Actual); Primary Completion 2005-04-06 (Actual); Study Completion 2005-04-20 (Actual)

PRIMARY OUTCOMES:
Prevention of PONV in the 24 hours following end of surgery; Tolerability | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Diemunsch P, Gan TJ, Philip BK, Girao MJ, Eberhart L, Irwin MG, Pueyo J, Chelly JE, Carides AD, Reiss T, Evans JK, Lawson FC; Aprepitant-PONV Protocol 091 International Study Group. Single-dose aprepitant vs ondansetron for the prevention of postoperative nausea and vomiting: a randomized, double-blind phase III trial in patients undergoing open abdominal surgery. Br J Anaesth. 2007 Aug;99(2):202-11. doi: 10.1093/bja/aem133. Epub 2007 May 30. PMID 17540667
- [Background] Diemunsch P, Apfel C, Gan TJ, Candiotti K, Philip BK, Chelly J, Carides AD, Evans JK, Ho TW, Reiss T. Preventing postoperative nausea and vomiting: post hoc analysis of pooled data from two randomized active-controlled trials of aprepitant. Curr Med Res Opin. 2007 Oct;23(10):2559-65. doi: 10.1185/030079907X233115. PMID 17845742
- [Background] Goveia MG, DiNubile MJ, Dallas MJ, Heaton PM, Kuter BJ; REST Study Team. Efficacy of pentavalent human-bovine (WC3) reassortant rotavirus vaccine based on breastfeeding frequency. Pediatr Infect Dis J. 2008 Jul;27(7):656-8. doi: 10.1097/INF.0b013e318168d29e. PMID 18520448
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/policies-perspectives.html